CLINICAL TRIAL: NCT04350255
Title: STEISURE - Trident II - A Registerbased Multicentric Prospective Study
Brief Title: A Register Based Prospective Study During Implementation of a New Cup
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Principal Investigator, Maziar Mohaddes Ardebili, Sahlgrenska University Hospital, Sweden, Sahlgrenska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEISURE - Trident II
Record Dates: First submitted 2020-04-08; First posted 2020-04-17 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Prospective
Keywords: Hip arthroplasty; Implant survival; Clinical outcome; X-ray; Implant Migration; Patient reported outcomes
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trident II Hemispherical cup (Stryker Orthopaedics) (Active Comparator): Total hip arthroplasty using non cemented Trident II Hemispherical acetabular cup
  Interventions: Device: Total hip arthroplasty
- Trident II Tritanium cup (Stryker Orthopaedics) (Active Comparator): Total hip arthroplasty using non cemented Trident II Tritanium acetabular cup
  Interventions: Device: Total hip arthroplasty

INTERVENTIONS:
Device: Total hip arthroplasty — Total hip arthroplasty with a Trident II hemispherical cup
Device: Total hip arthroplasty — Total hip arthroplasty with a Trident II Tritanium cup

SUMMARY:
In a prospective register-based study, we aim to evaluate the implant survival, clinical outcomes and X-ray findings by following a cohort of patients operated with the Trident II cup.

DETAILED DESCRIPTION:
Data will be collected from a cohort consisting of minimum 500 total hip arthroplasties. The patients will be recruited from multiple high volume centers in Sweden. To determine if there is evidence of inferiority as per benchmarking recommendations by The Orthopaedic Data Evaluation Panel the following parameters will be studied: Clinical parameters such as EQ-5D, Oxford Hip Score and Forgotten Joint Score, preoperative and after 1, 3, 6 and 10 years. Conventional radiography will be done preoperatively, postoperatively, 3, 6 and 10 years after total hip replacement. CTMA will be done postoperatively, 3 and 6 month and 2 years after total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip replacement
* Eligible for uncemented fixation of the acetabular component
* Suitable for one of the stem designs from Stryker Orthopaedics
* Accepts follow-up according to the study protocol

Exclusion Criteria:

* Difficulties to understand written information due to language problems or other reasons
* Use of augments needed
* Acute hip fracture
* Tumor in the hip joint

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Implant survival at 3 years | 3 years
  Kaplan Meier survival data, cup revision and risk of revision used as endpoints

SECONDARY OUTCOMES:
Implant migration measured with Computer Tomography Microanalysis in a subcohort of patients motion Analysis (CTMA) in a sub-cohort of patients | CTMA will be done postoperatively, 3 month and 6 months and 2 years after total hip replacement
  Using Computer Tomography Micro-motion Analysis (CTMA) to measure implant migration in a sub-cohort of patients
Implant survival at 10 years | 10 years
  Kaplan Meier survival data, cup revision and risk of revision used as endpoints
EQ-5D | 10 years
  Patient-reported generic health outcome measure
Plain radiographs in a sub-cohort of patients | 10 years
  Using plain radiographs to evaluate signs of loosening and implant position
Adverse events using the national patient register | 10 years
  ICD codes för surgical and medical adverse events following primary total hip arthroplasty, as defined by the National Board of Health and Welfare will be merged with data in the SHAR (The Swedish Hip Arthroplasty Register). This database includes mainly secondary care visits
Adverse events using the regional VEGA database | 10 years
  ICD (International Classification of Diseases) codes för surgical and medical adverse events following primary total hip arthroplasty, as defined by the National Board of Health and Welfare will be merged with data in the SHAR (The Swedish Hip Arthroplasty Register). This regional database includes all contacts (both within primary and secondary care) for patients living in the region of Western Sweden
Oxford Hip Score | 10 years
  Patient-reported hip specific outcome measure
Forgotten Joint Score | 10 years
  Patient-reported hip specific outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics, Mölndal, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to regulations associated with national registers in Sweden alla data will be presented on an aggregated level, individual patient data will not be shared.